CLINICAL TRIAL: NCT01269996
Title: JanUmet Before Insulin Lantus In Eastern Population Evaluation Program (JUBILEE) In Type 2 Diabetic Patients
Acronym: JUBILEE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2010.523
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; JUBILEE Study; Janumet; Lantus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Insulin Glargine; Metformin; Gliclazide; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin followed by gliclazide and protaphane (Active Comparator)
  Interventions: Drug: Janumet, Lantus; Drug: metformin, gliclazide, protaphane
- Janumet followed by Lantus insulin injection (Active Comparator)
  Interventions: Drug: Janumet, Lantus; Drug: metformin, gliclazide, protaphane

INTERVENTIONS:
Drug: Janumet, Lantus — In this multicentre, randomized, open-label prospective study. Recruited patients will be randomized to one of the two treatment groups. Treatment efficacy and safety in terms of HbA1c control and hypoglycemic events will be evaluated.
  Treatment groups:
  Group 1 - Metformin followed by Sulfonylurea (Gliclazide) and supplementary intermediate-acting insulin (Protaphane) injection.
  Group 2 - Janumet followed by Lantus insulin injection.
Drug: metformin, gliclazide, protaphane — In this multicentre, randomized, open-label prospective study. Recruited patients will be randomized to one of the two treatment groups. Treatment efficacy and safety in terms of HbA1c control and hypoglycemic events will be evaluated.
  Treatment groups:
  Group 1 - Metformin followed by Sulfonylurea (Gliclazide) and supplementary intermediate-acting insulin (Protaphane) injection.
  Group 2 - Janumet followed by Lantus insulin injection.

SUMMARY:
To evaluate the efficacy and safety of a new treatment regimen of metformin plus sitagliptin (Janumet) followed by a long-acting basal insulin (Lantus) treatment compared to the usual treatment regimen of metformin followed by sulfonylurea and intermediate-acting basal insulin in Type 2 Diabetes Mellitus patients.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) accounts for more than 90% of all diabetes. The worldwide prevalence of T2DM is increasing.

Microvascular and macrovascular complications are well known to cause significant morbidities and shorten life expectancy in diabetic patients. T2DM is the leading cause of adult-onset blindness, renal failure, limbs amputation, ischaemic heart disease and stroke in the industrialized world. Progressive pancreatic beta-cell failure together with insulin resistance underlie the pathogenesis of T2DM.

Glycaemic control is essential and fundamental to the management of diabetes. Randomized control trials have confirmed the long term benefits of achieving glycaemic control early in the course of disease on future clinical outcomes. Long term follow up of The Diabetes Control and Complications Trial Research Group (DCCT) and U.K. Prospective Diabetes Study (UKPDS) cohorts showed that improving glycaemic control reduces the incidences of both microvascular and macrovascular complications.

It is generally agreed that HbA1c <7% is a reasonable goal in adults to reduce risk of diabetes complications. Subgroup analyses of DCCT and UKPDS and results of Action in Diabetes and Vascular Disease: Preterax and Diamicron Modified Release Controlled Evaluation (ADVANCE) trial suggest a small but incremental benefit in microvascular outcomes with HbA1c values closer to normal. In the subgroup analysis of the ACCORD study, subjects without history of cardiovascular disease and attained HbA1c goal of 6.5% had lower risk of cardiovascular endpoints than those with HbA1c goal of 7%. Therefore, selected individual patients including those with short duration of diabetes, long life expectancy and no significant cardiovascular disease, may benefit from a more stringent HbA1c goal of <6.5%, a value close to normal individual.

According to the American Diabetes Association (ADA) and the European Association for the Study of Diabetes, lifestyle modification plus Metformin is a well-validated step 1 therapy for patients with T2DM. Sulfonylurea or insulin treatment formed the step 2 therapy in those who fail to achieve optimal glycaemic control after step 1 treatment. Sulfonylurea is an insulin secretagogue. It acts in a glucose-independent fashion by increasing the insulin concentration irrespective of the ambient glucose concentration. Despite its efficacy, it is associated with increased risk of hypoglycaemia and weight gain.

Incretins are gut-derived hormones that include Glucagon-like peptide-1 (GLP-1) and Glucose-dependent insulinotropic peptide (GIP). Incretins are released into the circulation after a meal. Both GLP-1 and GIP stimulate endogenous insulin secretion in a glucose-dependent fashion. They also inhibit glucagon secretion, delay gastric emptying and induce satiety. The combined effect of incretins in augmenting insulin secretion and suppressing glucagon reduces post-prandial glucose excursion. In animal models, GLP-1 has also been shown to preserve pancreatic beta-cell mass by increased proliferation and decreased apoptosis. In T2DM patients, the attenuated post-prandial GLP-1 secretion may partially explain the increased post-prandial rise in glucose concentration.

However, incretins have very short half-lives of a few minutes. They are rapidly inactivated by the enzyme dipeptidyl peptidase IV (DPP-4) in the circulation. Inhibitors of the enzyme DPP-4 can augment active incretin levels by delaying the clearance of the active incretins, hence augmenting the incretin action with resultant improvement in glycaemic control in T2DM patients.

In later stage of T2DM, progressive pancreatic beta-cell failure frequently results in deterioration in glycaemic control despite oral drug treatment, necessitating supplementary insulin therapy. New generations of once-daily, long-acting basal insulin may have better safety profile in terms of less hypoglycaemic events compared with traditional intermediate-acting basal insulin. Supplementary basal insulin, when titrated appropriately, will almost always improve fasting blood glucose levels and HbA1c control.

Sitagliptin is an orally active, potent and highly selective DPP-4 inhibitor which was approved by the U.S. Food and Drug Administration (FDA) in October 2006 as a new class of oral drug treatment for T2DM. Sitagliptin is marketed as Januvia by Merck & Co. In April 2007, the FDA approved an oral combination of sitagliptin and metformin marketed as Janumet with preparations of 50/500mg and 50/1000mg dosage per tablet. Sitagliptin has been proved to be effective in treating T2DM with minimal risk of hypoglycaemia together with additional benefits on reducing glucagon, slowing gastric emptying and inducing satiety.

Insulin glargine, marketed by Sanofi Aventis under the name Lantus, is a long-acting basal insulin analogue. It has the advantage of a long action duration of 18 to 26 hours and a peakless profile, which resembles basal insulin secretion of non-diabetic pancreatic beta-cells.

In T2DM patients, we proposed that a new treatment regimen consists of a combination of DPP-IV inhibitor plus metformin followed by long-acting basal insulin may be more effective in achieving good and sustained glycaemic control with less hypoglycaemic drawbacks compared with the traditional regimen of metformin followed by sulfonylurea and finally intermediate-acting insulin. This proposed new treatment regimen forms the basis of this study.

The objective of this multicentre, randomized, open-label prospective study is to evaluate the efficacy and safety of a new treatment regimen of metformin plus sitagliptin (Janumet) followed by a long-acting basal insulin (Lantus) treatment compared to the usual treatment regimen of metformin follow by sulfonylurea and intermediate-acting basal insulin in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 to 80 years old at Visit 1.
2. Male or female of Chinese ethnicity.
3. Type 2 diabetic patients who are drug naïve with HbA1c ranged between 7.0% to 11.0%.
4. Type 2 diabetic patients who are on single oral hypoglycaemic drug treatment or insulin treatment of duration less than 6 months are eligible after at least 3 months of washout period with diet control only prior to Visit 1 and satisfy the inclusion criteria of HbA1c ranged between 7.0% to 11.0%.
5. Patient understands the study procedures, alternative treatments available, and the risks involved with the study, and voluntarily agrees to participate by providing written informed consent.
6. Patient agrees to provide permission to obtain all medical records necessary for complete data ascertainment during study and follow-up period.

Exclusion Criteria:

1. Patient has a history of type 1 diabetes mellitus or a history of ketoacidosis.
2. Patients with HbA1c 9% to 11% who have severe symptoms and showing signs of decompensation (e.g. rapid weight loss and ketonuria) due to hyperglycaemia.
3. On anti-obesity drugs 12 weeks prior to informed consent, patient in a weight loss program or intends to be involved in weight loss intervention outside that prescribed by the study.
4. Patient has renal impairment defined as serum creatinine equal to/more than 123 umol/l (1.4mg/dL) in female and serum creatinine equal to/more than 132 umol/l (1.5mg/dL) in male.
5. Significant liver impairment (ALT equal to /more than 2 times upper limit of normal range) or a medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, liver cirrhosis or symptomatic gallbladder disease.
6. Any history of cardiovascular disease, stroke or peripheral vascular disease.
7. Any symptoms of ischaemic heart disease like angina.
8. Renal transplant patients.
9. Active malignant disease. Patients with malignant disease who have been successfully treated and disease-free for at least 5 years are eligible. However, patients with a history of leukaemia, lymphoma, aplastic anaemia, myeloproliferative or myelodysplastic disease, thrombocytopenia, malignant melanoma, or renal cell carcinoma are ineligible for the study regardless of the time since treatment.
10. Patient has medical history that indicates a life expectancy of less than 5 years or might limit the individual's ability to take trial treatments for the duration of the study.
11. Patient has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance which, in the opinion of the investigator or coordinator, might pose a risk to the patient, make participation not in the patient's best interest, confound the results of the study (e.g. if patient cannot comply with requirements of the study), or interfere with the patient's participation for the full duration of the study.
12. Patient has a known history of hypersensitivity, intolerance or any contraindication to either metformin, sulfonylurea, DPP-IV inhibitor or insulin.
13. Active and uncontrolled thyroid diseases or active endocrine diseases like Cushing's syndrome or acromegaly.
14. Pre-menopausal women (last menstruation 1 year prior to signing informed consent) who: are nursing or pregnant, or are of child-bearing potential and are not practicing an acceptable and reliable contraceptive methods, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intra-uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner. No exception will be made.
15. Any medical illness or condition as judged by the investigators as ineligible to participate the study.
16. Special population, e.g. prisoner, mentally disabled, persons with psychiatric disorders and investigators' student or employees.
17. Patient is currently participating in or has participated in another study with an investigational compound or device within the prior 12 weeks of screening or signing the informed consent and does not agree to refrain from participating in any other study while participating in this study.
18. Patient has undergone surgery within the prior 12 weeks or has major surgery planned during the study.
19. Patient is on or is likely to require treatment with equal to/ more than 14 consecutive days or repeated courses of pharmacologic doses of corticosteroids.

    Note: Inhaled, nasal, and topical corticosteroids are permitted.
20. Patient has a clinically significant laboratory or ECG abnormality which, in the opinion of the investigator, exposes the patient to risk by enrolling in the study.
21. History of drug abuse or alcohol abuse. History of recreational or illicit drugs used. Alcohol abuse includes heavy alcohol intake as defined by more than 2 drinks per day or more than 14 drinks per week, or binge drinking.
22. Patient has a clinically significant haematological disorder (e.g., aplastic anaemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia, thalassaemia or thalassaemia trait).
23. Blood donation 3 months prior to the start of the study and during the whole study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-05; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the treatment efficacy | one year
  The change in HbA1c in 1 year compare to baseline.

SECONDARY OUTCOMES:
proportion of patients with HbA1c <6.5% in 1 year | one year
  Secondary Outcome Measure: The proportion of patients with HbA1c <6.5% in 1 year.
  Other outcome measures: a)The change in body weight compare to baseline. b)Frequency of hypoglycaemia . Hypoglycemia is defined according to the ADA definitions and classifications of hypoglycaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana CN CHAN, FRCP, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong